## Version 1.1 Version date 02/07/2019

## CONSENT BY PATIENT FOR CLINICAL RESEARCH

| I, |
|---|
| of |
| (Address) hereby agree to take part in the clinical research (clinical study/questionnaire study/drug trial) specified below: |
| <u>Title of Study:</u> The Effect of 30-Minute Mindful Breathing in Reducing Fatigue Symptom among Patients |
| with Haematological Cancer – A Randomized Controlled Trial. |
| the nature and purpose of which has been explained to me by Dr |
| (Name & Designation of Doctor) |
| and interpreted by |
| (Name & Designation of Interpreter) |
| to the best of his/her ability in |
| I have been told about the nature of the clinical research in terms of methodology, possible adverse effects and complications (as per patient information sheet). After knowing and understanding all the possible advantages and disadvantages of this clinical research, I voluntarily consent of my own free will to participate in the clinical research specified above. |
| I understand that I can withdraw from this clinical research at any time without assigning any reason whatsoever and in such a situation shall not be denied the benefits of usual treatment by the attending doctors. |
| Date: Signature or Thumbprint |
| (Patient) |
| IN THE PRESENCE OF |
| Name) |
| Identity Card No |
| (Witness for Signature of Patient) |
| Designation) |
| I confirm that I have explained to the patient the nature and purpose of the above-mentioned clinical research. |
| Date |

CONSENT BY PATIENT FOR CLINICAL RESEARCH

R.N. Name Sex Age Unit

BK-MIS-1117-

## Version 1.1 Version date 02/07/2019

## CONSENT BY RESPONSIBLE RELATIVE FOR CLINICAL RESEARCH

| I, | | |
|---|---|---|
| Identity Card No(Name) | | |
| of | | |
| (Address) | | |
| hereby agree that my relative | stionnaire study/drug trial) | |
| Patients with Haematological Cancer - A Randomiz | ed Controlled Trial. | |
| the nature and purpose of which has been explained | to me by Dr. | |
| (Name & Designation of Doctor) | | |
| and interpreted by(Name & Designation of Inter | | |
| to the best of his/her a | bility in | language/dialect. |
| I have been informed of the nature of this clinical reand complications (as per patient information sidisadvantages of participating in this research. I volin this research specified above. | heet). I understand the | possible advantages and |
| I understand that I can withdraw my relative from the reason whatsoever and in such situation, my relative the attending doctors. Should my relative regains he remain in this research or may choose to withdraw. | shall not be denied the bene | efits of usual treatment by |
| Relationship Date: to Patient | Signature or<br>Thumbprint | |
| IN THE PRESENCE OF | | |
| Name) | | |
| Identity Card No) | Signature | (Witness) |
| Designation | | ` |
| I confirm that I have explained to the patient's relatively clinical research. | e the nature and purpose of | f the above-mentioned |
| Date | Signature | |
| | (Attending Doctor | r) |